CLINICAL TRIAL: NCT02191683
Title: Foetal Exposure and Epidemiological Transition: the Role of Anaemia in Early Life for Non-communicable Diseases in Later Life
Brief Title: Foetal Exposure and Epidemiological Transition: Role of Anaemia in Early Life for Non-communicable Diseases Later
Acronym: FOETALforNCD
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Copenhagen University Hospital, Denmark (Other); Aarhus University Hospital (Other); Lund University (Other); National Institute for Medical Research, Tanzania (Other Government); Department of Clinical Pathology Naestved Hospital Denmark (Unknown)
Responsible Party: Principal Investigator, Ib Christian Bygbjerg, Professor, University of Copenhagen
Other Study IDs: 1309-00003B; Strategiske Forskningsråd (Other: Danish Council for Strategic Research)
Record Dates: First submitted 2014-07-02; First posted 2014-07-16 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Anemia and Pregnancy; Metabolism and Foetal Growth; Epigenetics
Keywords: Anaemia; Pregnancy; Foetal programming; Epigenetics; Non-communicable diseases; Tanzania
MeSH Terms: conditions — Anemia; Noncommunicable Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Months
Biospecimen Retention: Samples With DNA — Periperal vein blood, umbilical cord blood, placentas
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Health of women before conception: Tanzanian women aged 18-40 years focusing on prevalence of anaemia, infections, nutritional status, and NCDs.
- 480 women during pregnancy: Describe how 1st and 2nd trimester anaemia compared to 3rd trimester anaemia alters foetal growth and newborns' body composition.
  Evaluate anaemia's effect on villous branching in placenta, and uterine and umbilical artery blood flow.
  Evaluate effect on vascular endothelial growth factor A/placental growth factor balance and insulin-like growth factor axis.
  Determine which markers for foetal programming such as methylation of regulatory genes related to metabolism and haematopoiesis may be discovered early after exposure to anaemia.

SUMMARY:
Study Hypotheses:

1. Anaemia, which is frequent before conception as well as during early pregnancy, affects metabolism and foetal growth trajectories, influencing the risk of NCDs in the offspring.
2. Anaemia from conception till end of 2nd trimester is most detrimental for foetal and newborns' health, compared to 3rd trimester anaemia.
3. Anaemia from conception till end of 2nd trimester affects foetal and newborns health through poor placental development reflected in increased villous branching and changed umbilical and uterine blood flow.
4. Anaemia in early pregnancy disrupts the vascular endothelial growth factor A (VEGF-A)/placental growth factor (PlGF) balance and the insulin-like growth factor (IGF) axis resulting in poor placental development, and poor health of newborns. This may be reflected in specific methylation patterns.
5. Anaemia's impact on the risk for NCDs in the offspring may be mediated via epigenetic mechanisms, including changes in DNA methylation patterns.

DETAILED DESCRIPTION:
Specific objectives are:

1. Characterize the health of women aged 18-40 years before conception and during pregnancy, focusing on prevalence of anaemia, infections, nutritional status, and Non-Communicable Diseases (NCDs).
2. Describe how 1st and 2nd trimester anaemia compared to 3rd trimester anaemia alters foetal growth and newborns' body composition.
3. Evaluate how 1st and 2nd trimester anaemia compared to 3rd trimester anaemia affects villous branching in the placenta, as well as uterine and umbilical artery blood flow.
4. Characterize how 1st, 2nd and 3rd trimester anaemia differentially changes the vascular endothelial growth factor A (VEGF-A)/placental growth factor (PlGF) balance and the insulin-like growth factor axis.
5. Determine which markers for foetal programming such as methylation of regulatory genes related to metabolism and haematopoiesis may be discovered early after exposure to anaemia in1st and 2nd trimester compared to 3rd trimester anaemia.

Outcome parameter for the pre-pregnancy study (i.): 1) Prevalence and severity of anaemia among non-pregnant Tanzanian women at fertile age and their nutritional status. 2) Incidence of conception among such women.

Outcome parameter for the pregnancy study (ii.): 1) Foetal growth rate in 2nd and 3rd trimester in offspring of anaemic mothers vs Foetal growth rate in non-anaemic mothers' offspring, 2) Comparison of anaemic mothers' vs non-anaemic mothers' newborn's body composition, placental villous branching, umbilical and uterine blood flow, VEGF-A/PlGF levels, and insulin-like growth factor axis.

For all analyses main exposure variable will be anaemia (Hb<5mmol/L) in 1st, 2nd and/or3rd trimester of pregnancy. Confounding exposure variables will be chronic health conditions (e.g. HIV), all temporary conditions mentioned above (e.g. malaria) as well as socioeconomic status and paternal characteristics. Regression modelling using both multiple linear and logistic regressions as well as modelling for repeated measures will be used for statistical analyses. For genetic and epigenetic changes, findings in the subgroup of 180 other/newborns, remaining significant after correction for multiple comparisons, will be validated in the remaining cohort. This will enable us within one study to replicate initial findings in one representative and distinct subgroup in another larger comparable study group from an overall homogenous study. Indeed, findings surviving both corrections for multiple testing in the initial hypothesis generating array approaches, as well as being replicated in the remaining study group with single target validation techniques, are highly likely to be biological important. Possible findings from the candidate gene approach will be corrected for multiple testing and the significant results will be compared with previous findings of the same genes from studies in muscle and adipose tissue conducted by Diabetes and Metabolism, Copenhagen University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* wishing to get pregnant
* negative pregnancy test
* not using family planning

Exclusion Criteria:

* not wishing to get pregnant
* being pregnant
* using family planning

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Amendment October 2014: replacement of two-phase case-control study by two sub-projects, running in parallel, and following two distinct groups of women, 1) a cohort of 1500 non-pregnant women, disregarding Hb level, of whom 270 followed throughout pregnancy disregarding Hb level and gestational age at first contact, and 2) a case control study of 480 pregnant women followed from 1st trimester with a 160:160:160 ratio of women with Hb≤8g/dL: 8.1-10.9g/dL: ≥11g/dL.
  The Danish Council for Strategic Research notified and accepted in November 2014.
Sampling Method: Probability Sample
Enrollment: 1748 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Outcome parameter for the pre-pregnancy study (i.): | 12 months from start
  Prevalence and severity of anaemia among non-pregnant Tanzanian women at fertile age and their nutritional status.
Outcome parameter for the pregnancy study (ii.): | 31 months
  Anemia's effect on foetal growth rate in 2nd and 3rd trimester measured as a) discrepancy in estimated and predicted gestational age (GA) between inclusion and antenatal visit at GA 20 weeks & 30, b) change in z-score for foetal weight/body weight and c) gain in g/week26 at GA of 26, 32 and 37 and delivery. Newborn's body composition, placental villous branching, umbilical and uterine blood flow, VEGF-A/PlGF levels, and GFaxis. For all analyses main exposure variable are anaemia in 1st, 2nd and/or3rd trimester of pregnancy. Confounding exposure variables are chronic health conditions, temporary conditions mentioned above (e.g. malaria) and socioeconomic status and paternal characteristics. Regression modelling using multiple linear and logistic regressions and modelling for repeated measures are used for statistical analyses. Genetic and epigenetic significant changes in subgroup of 180 mother/newborns, after correction for multiple comparisons, will be validated in remaining cohort.
Incidence of conception among non-pregnant Tanzanian women. | 12 months
  Number of women screened, with and without anaemia, respectively, who actually become pregnant within the observation period

CONTACTS AND LOCATIONS:
Overall Officials: Mwelecele N Malecela, PHd, Study Chair — National Institute for Medical Research, Tanzania
Locations (1):
- National Institute for Medical research, Korogwe, Tanga, Tanzania

REFERENCES:
- [Derived] Hatem G, Hjort L, Asplund O, Minja DTR, Msemo OA, Moller SL, Lavstsen T, Groth-Grunnet L, Lusingu JPA, Hansson O, Christensen DL, Vaag AA, Artner I, Theander T, Groop L, Schmiegelow C, Bygbjerg IC, Prasad RB. Mapping the Cord Blood Transcriptome of Pregnancies Affected by Early Maternal Anemia to Identify Signatures of Fetal Programming. J Clin Endocrinol Metab. 2022 Apr 19;107(5):1303-1316. doi: 10.1210/clinem/dgac010. PMID 35021220
- [Derived] Paulsen CB, Nielsen BB, Msemo OA, Moller SL, Ekmann JR, Theander TG, Bygbjerg IC, Lusingu JPA, Minja DTR, Schmiegelow C. Anthropometric measurements can identify small for gestational age newborns: a cohort study in rural Tanzania. BMC Pediatr. 2019 Apr 23;19(1):120. doi: 10.1186/s12887-019-1500-0. PMID 31014291
- [Derived] Moeller SL, Nyengaard JR, Larsen LG, Nielsen K, Bygbjerg IC, Msemo OA, Lusingu JPA, Minja DTR, Theander TG, Schmiegelow C. Malaria in Early Pregnancy and the Development of the Placental Vasculature. J Infect Dis. 2019 Sep 26;220(9):1425-1434. doi: 10.1093/infdis/jiy735. PMID 30590576
- [Derived] Msemo OA, Bygbjerg IC, Moller SL, Nielsen BB, Odum L, Perslev K, Lusingu JPA, Kavishe RA, Minja DTR, Schmiegelow C. Prevalence and risk factors of preconception anemia: A community based cross sectional study of rural women of reproductive age in northeastern Tanzania. PLoS One. 2018 Dec 18;13(12):e0208413. doi: 10.1371/journal.pone.0208413. eCollection 2018. PMID 30562390